CLINICAL TRIAL: NCT03228914
Title: Comparing Blood Loss and Visualization After the Preoperative Use of Topical 0.05% Oxymetazoline Versus 1:1000 Epinephrine Prior to Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, William Yao, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-17-0415
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Endoscopic Sinus Surgery; Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Oxymetazoline; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxymetazoline (Active Comparator): Pledgets will be soaked in 0.05% oxymetazoline solution Two pledgets with the associated medication will be placed into the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
  Interventions: Drug: Oxymetazoline
- Epinephrine (Active Comparator): Pledgets will be soaked in 1:1000 epinephrine solution Two pledgets with the associated medication will be placed into the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Oxymetazoline — Pledgets will be soaked in 0.05% oxymetazoline solution Two pledgets with the associated medication will be placed into the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
  Other Names: Afrin
  Arms: Oxymetazoline
Drug: Epinephrine — Pledgets will be soaked in 1:1000 epinephrine solution Two pledgets with the associated medication will be placed into the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
  Arms: Epinephrine

SUMMARY:
The purpose of this study is to compare the effects of Oxymetazoline and Epinephrine (which are 2 different nasal decongestants both of which are routinely used before sinus surgery) on blood loss and the surgeon's view of the surgical field during sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be patients undergoing bilateral endoscopic sinus surgery (ESS) in which the same sinuses and procedures on both sides are the same for CRS with or without nasal polyposis.

Exclusion Criteria:

* pregnancy
* known coagulopathy
* an international normalized ratio greater than 1.3
* a partial thromboplastin time greater than 50 seconds
* use of non-steroidal anti-inflammatory drugs in the last 10 days (2 or more doses)
* use of any antiplatelet agents (eg, warfarin, clopidogrel, berlinta)
* poorly controlled hypertension with a preoperative systolic blood pressure of 160mm Hg or greater or a diastolic blood pressure of 90mm Hg or greater
* having any adverse reaction to topical epinephrine or oxymetazoline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Yao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For each participant who started the study, oxymetazoline was administered to one side of the nasal cavity and epinephrine was administered to the other side of the nasal cavity. Each participant has two sides of the nasal cavity, and each participant received both oxymetazoline and epinephrine, one drug per side.
Units Other Than Participants: one side of nasal cavity
Period: Overall Study
Arm/Group | Oxymetazoline | Epinephrine
Started | 20; 20 one side of nasal cavity | 20; 20 one side of nasal cavity
Completed | 20; 20 one side of nasal cavity | 20; 20 one side of nasal cavity
Not Completed | 0; 0 one side of nasal cavity | 0; 0 one side of nasal cavity

BASELINE CHARACTERISTICS:
Population: Adults greater than 18 years of age undergoing endoscopic sinus surgery. Age is an inclusion criteria and is not collected
Groups:
- All Participants: Pledgets will be soaked in 0.05% oxymetazoline solution Two pledgets with the associated medication will be placed into one side of the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
  Pledgets will be soaked in 1:1000 epinephrine solution Two pledgets with the associated medication will be placed into the other side of the nasal cavity; one along the floor of the nose and another directed towards the middle meatus.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data were not collected as part of the study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Presence of polyps [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Surgical Field Visualization During Sinus Surgery as Indicated by Score on Boezaart Grading Scale
Description: The minimum Boezaart Grading Scale score of 0 indicates no bleeding (cadaveric conditions), and the maximum score of 5 indicates severe bleeding (constant suctioning required).
Time Frame: during surgery approximately 2-3 hours
Population: For each participant who started the study, oxymetazoline was administered to one side of the nasal cavity and epinephrine was administered to the other side of the nasal cavity. Each participant has two sides of the nasal cavity, and each participant received both oxymetazoline and epinephrine, one drug per side.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: one side of nasal cavity
Arm/Group | Oxymetazoline | Epinephrine
Number analyzed (Participants) | 20 | 20
Number analyzed (one side of nasal cavity) | 20 | 20
score on a scale | 3 (0.19) | 2.55 (0.15)

2. Secondary Outcome: Amount of Blood Loss in mL
Description: The secondary endpoint will be to compare the amount of blood loss use after the use of epinephrine or Oxymetazoline. This will be done by subtracting the amount of irrigation used from the volume collected in the suction canisters to estimate blood loss. The Neptune 2 Waste Management System (NWMS, Stryker, Kalamazoo, Michigan), a closed suction system that digitally measures the amount of fluid suctioned will be used for more accurate measuring of fluid suctioned. Surgery lasts about 2-3 hours, and the suctioning stops immediately following the completion of the case.
Time Frame: immediately at the completion of surgery (surgery lasts about 2-3 hours, and the suctioning stops immediately following the completion of the case)
Population: Data was not collected for this measure.
Arm/Group | Oxymetazoline | Epinephrine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse event was collected during the surgical case on the day the patient was enrolled. (2-3hours)
Description: Adverse events were collected if there were any deviations to the surgery or patients hemodynamic status while using the pledgets.
Arm/Group | Oxymetazoline | Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03228914/Prot_SAP_000.pdf